CLINICAL TRIAL: NCT04973371
Title: Investigating the Acceptability and Feasibility of Home-based TB Testing of Household Contacts Using a New, Mobile Point-of-care Technology
Brief Title: Acceptability and Feasibility of Home-based TB Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Professional Development (Pty) Ltd (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Medical Research Council, South Africa (Other); Foundation for Innovative New Diagnostics, Switzerland (Other); University of Witwatersrand, South Africa (Other); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R21EB023679 (NIH); R21EB023679 (NIH)
Record Dates: First submitted 2021-06-30; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Tuberculosis, Pulmonary; Households
Keywords: Tuberculosis; Household Contacts; Household Contact Investigation; Active Case Finding; Home-based Testing; GeneXpert; Point-of-Care Testing; South Africa; Tuberculosis symptomatic household contacts
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Intervention Model Description: An exploratory study to 1) investigate the acceptability and feasibility of home-based TB testing of household contacts using a new portable GeneXpert point-of-care (PoC) platform, and 2) determine the potential impact of such a home-based testing program on early detection of TB disease and linkage-to-care (LTC). In this study, all participants enrolled in the Treatment arm will be tested for TB at their household, using the GeneXpert device. Participants enrolled in the Control arm will receive a referral letter, which can be used to access treatment at the nearest health facility. No single participant will be randomized, the whole house will receive a "Blanket Randomisation".
Masking Description: The allocation of study arm is concealed to study staff during randomization. Neither study staff nor participants will be blinded to study treatment arms after the point of randomization. Nonetheless, strict policies will be in place to preserve randomization integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based GeneXpert TB test (Experimental): Screening household contacts + home-based GeneXpert® MTB/RIF TB testing for those with TB symptoms + immediate referral for clinic-based treatment initiation.
  Interventions: Diagnostic Test: Home-based point-of-care (POC) TB testing using GeneXpert device + MTB/RIF test
- Standard home-based TB symptom screening with immediate referral (No Intervention): Screening household contacts + immediate referral for clinic-based TB testing

INTERVENTIONS:
Diagnostic Test: Home-based point-of-care (POC) TB testing using GeneXpert device + MTB/RIF test — Those who screen positive for TB using the standard 4-question screener will be offered a GeneXpert® [Cepheid, Sunnyvale, CA] MTB/RIF test in their home with referral for clinic-based TB treatment initiation for those who receive a positive MTB/RIF test result.
  Arms: Home-based GeneXpert TB test

SUMMARY:
This study aims to evaluate the utility of home-based point-of-care TB testing for early diagnosis and linkage to care of household contacts of TB patients, addressing the need for active case finding and early detection of infectious TB. The investigators propose an exploratory study to 1) investigate the acceptability and feasibility of home-based TB testing of household contacts using a new portable GeneXpert point-of-care (PoC) platform, and 2) determine the potential impact of such a home-based testing program on early detection of TB disease and linkage-to-care (LTC).

DETAILED DESCRIPTION:
In 2013, WHO estimated that 3.3 million cases of TB had been missed (undiagnosed or with a significant delay in diagnosis or treatment). "Missed" TB cases are a key driver of TB transmission, with approximately 9 million individuals developing TB globally each year, equivalent to 126 cases per 100,000 population. The overall goal of this proposal is to evaluate the utility of home-based point-of-care TB testing for early diagnosis and linkage to care of household contacts of TB patients, addressing the need for intensive case finding and early detection of infectious TB. Although well-accepted as an effective strategy for boosting HIV diagnosis and treatment rates, until recently home-based testing for TB has been impossible, as there has never existed an effective, mobile PoC technology for rapid diagnosis of TB. With the development of the new GeneXpert® Omni diagnostic platform from Cepheid, home-based TB testing is now possible. Now is the time to study whether home-based testing for TB is feasible, and will contribute to early case detection or improve time-to-treatment rates.

This project has two Specific Aims:

1. To determine the acceptability and feasibility of using point-of-care technology to perform home-based TB testing of household contacts of TB patients, with subaim 1(a): To assess the intent-to-seek care of household contacts symptomatic for TB, and subaim 1(b): To determine the proportion of household contacts symptomatic for TB consenting to be tested (acceptability) and uptake of treatment referrals by those individuals infected with TB within 30 days of testing (feasibility);
2. To describe the outcomes of household contacts screened and tested for TB in their home compared to those screened and referred for testing in a health facility, with subaim 2(a): To describe the barriers and facilitators to clinic follow-up by household contacts symptomatic for TB and provided with referral for TB testing or treatment initiation, and subaim 2(b): To determine whether point-of-care home-based TB testing reduces time-to-treatment initiation.

An exploratory study will be conducted in a high TB prevalence area of Eastern Cape Province, South Africa. Specifically, households of TB patients initiating treatment at one of 6 collaborating clinics will be offered a point-of-care home-based TB test, with referral for immediate treatment when testing positive. In accordance with the South African National TB Management Guidelines (SA-NTMG), all smear positive pulmonary TB (PTB) patients recruited and consented will be asked to provide a list of all household contacts for a household contact investigation. The household contact investigation team will then, in keeping with South African National Department of Health guidelines, seek verbal consent from all household contacts to conduct TB symptom screening. During symptom screening, intent-to-seek care will be assessed for all reported symptoms. If one household member screens positive, then the whole household will be randomized to either the Intervention; home-based GeneXpert point-of-care (PoC) test or Control arm; standard home-based TB symptom screening with referral for testing.

ELIGIBILITY:
Inclusion Criteria:

* TB symptomatic household contact of a TB patient
* Not currently on TB treatment
* Able to produce a sputum specimen for testing
* Age ≥18 years
* Provision of written consent

Exclusion criteria

* Unable to speak and answer questions in English, Xhosa or Afrikaans
* Household contact has already been to the facility for TB testing or is already on TB treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of home-based TB testing | Within 1 hour
  ≥ 80% of individuals who screen positive for TB consent to home-based testing using the GeneXpert Platform.
Feasibility of home-based TB testing | Within 1 hour
  ≥80% of households visited having a safe space for sputum production. A safe space for sputum production and collection will be defined as per the South African 2014 National TB Management Guidelines.
Feasibility of home-based TB testing | Immediate upon test completion
  >90% of MTB/Rif tests produce a valid test result
Feasibility of home-based TB testing | Within 4 weeks of diagnosis
  ≥ 80% of household contacts testing positive for TB present at a clinic for care and treatment

SECONDARY OUTCOMES:
Proportion of referral uptake | Within 30 days
  Proportion of household contacts presenting for clinical follow up. (Number of household contacts presenting for clinical follow up / total household contacts referred for clinical follow-up)
Time to clinic presentation | Within 30 days
  Number of days elapsed between date of household contact investigation and date of initial presentation to the clinic.
Time-to-treatment initiation | Within 30 days
  Number of days elapsed between date of household contact investigation and date of TB treatment initiation.
Proportion initiating treatment | Within 30 days
  Number household contacts diagnosed with TB initiating treatment / total household contacts diagnosed with TB

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Medina-Marino, PhD, Principal Investigator — andrewmedinamarino@gmail.com
Locations (1):
- Buffalo City Metro, East London, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on public repository 1) in parallel with manuscript publication or 2) within two years of study completion (whichever comes earlier)
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Supporting information will be made available as requested 1) in parallel with manuscript publication or 2) within two years of study completion (whichever comes earlier)